CLINICAL TRIAL: NCT04189432
Title: A Multicenter, Randomized, Parallel Group, Double-blind, Phase 2 Trial to Evaluate Efficacy and Safety of SCM-CGH in Patients With Steroid-Refractory or Dependent Chronic Graft-Versus-Host Disease
Brief Title: Efficacy and Safety of SCM-CGH in Patients With Steroid-Refractory or Dependent Chronic Graft-Versus-Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SCM Lifescience Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCM-CGH2001
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Chronic Graft-versus-host-disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: A Multicenter, Randomized, Parallel Group, Double-blind
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCM-CGH (Experimental): * Ingredient: Allogeneic human bone marrow-derived mesenchymal stem cells
  * Dose: 1x10^6 cells/Kg
  Interventions: Biological: SCM-CGH
- Placebo (Placebo Comparator): 3 times with 2-week intervals by IV infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: SCM-CGH — SCM-CGH will be administrated 3 times with 2-week intervals by IV infusion to subjects at Weeks 0, 2 and 4 (Visits 2, 3 and 4).
  Arms: SCM-CGH
Other: Placebo — Placebo will be administrated 3 times with 2-week intervals by IV infusion to subjects at Weeks 0, 2 and 4 (Visits 2, 3 and 4).
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy of SCM-CGH in participants with steroid dependent/refractory chronic graft versus host disease (cGVHD) by measuring overall cGVHD response (complete response [CR] and partial response [PR] defined by National Institutes of Health [NIH] consensus development project criteria [2014]).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are males or females aged >= 19 years, 40kg to 80kg in weight
* Steroid dependent/refractory chronic graft versus host disease (cGVHD) defined as the National Institutes of Health (NIH) criteria (2014) below at any time post-hematopoietic cell transplant (post-HCT):

Refractory disease, defined as, 1) when cGVHD manifestations progress despite the use of a regimen containing glucocorticoid (prednisolone at >=1 mg/kg/day for at least 2 weeks) or 2), 3) Persist without improvement despite continued treatment with glucocorticoid (prednisolone at >=0.5 mg/kg/day or 1 mg/kg every other day) for at least 4 weeks Dependent disease, defined as, 4), 5) when glucocorticoid (prednisolone doses greater than or equal to [>=] 0.25 milligram per kilogram per day (mg/kg/day)or >=0.5 milligram per kilogram (mg/kg) every other day) are needed to prevent recurrence or progression of manifestations as demonstrated by unsuccessful attempts to taper the dose to lower levels on at least 2 occasions, separated by at least 8 weeks.

* Participants must be receiving less than 3 systemic glucocorticoid therapies or other immunosuppressive therapies in addition to glucocorticoids for cGVHD for at least 4 weeks before Screening visit. The dose of steroids or Immunosuppressant must be stable for 14 days(2 weeks) prior to starting SCM-CGH or Placebo.
* Laboratory test sufficiency as follows; Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3 Serum creatinine < 2 x upper limit of normal (ULN)

Exclusion Criteria:

* Active acute graft versus host disease (GVHD)
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus (HCV)
* Uncontrolled underlying disease such as moderate or severe infections and hemorrhage
* Severe Heart failure (NYHA class III/IV), congestive heart failure or arrhythmia requiring treatment
* History of allogenic hematopoietic stem cell more than once
* Positive reaction of a Penicillin test at screening
* History of relapse of causative diseases (ALL, CML, CLL, AML, NHL, multiple myeloma e.t.c.) with hematopoietic stem cell transplantation or diagnosed with secondary malignant diseases after hematopoietic stem cell transplantation
* History of Anti-thymocyte globulin(ATG) for 2 weeks before Screening visit
* History of pulmonary embolism or deep venous thrombosis for 24 weeks before Screening visit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-09-28 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve Complete Response (CR) or Partial Response (PR) (i.e. Overall Response Rate [ORR]) | Week 12
  ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR). Response is defined by the National Institutes of Health (NIH) Consensus Development Project Criteria (2014) and must occur, in the absence of new therapy for chronic graft versus host disease (cGVHD) and absence of progression of underlying disease or death. CR: Resolution of all manifestations in each organ or site. PR: Improvement in at least 1 organ or site without progression in any other organ or site. cGVHD Progression: Clinically meaningful worsening in 1 or more organs regardless of improvement in other organs.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve Complete Response (CR) or Partial Response (PR) (i.e. Overall Response Rate [ORR]). | Week 0, 2, 4, 6, 8, 16, 20, 24 and 48
  ORR is defined as the percentage of participants who achieve complete response (CR) or partial response (PR). Response is defined by the National Institutes of Health (NIH) Consensus Development Project Criteria (2014) and must occur, in the absence of new therapy for chronic graft versus host disease (cGVHD) and absence of progression of underlying disease or death. CR: Resolution of all manifestations in each organ or site. PR: Improvement in at least 1 organ or site without progression in any other organ or site. cGVHD Progression: Clinically meaningful worsening in 1 or more organs regardless of improvement in other organs.
Organ-specific Assessments | Week 0, 2, 4, 6, 8, 16, 20, 24 and 48
  Percentage of participants with organ-specific assessments is defined as rate of NIH defined CR or PR.
Patient-Reported Outcomes | Week 0, 2, 4, 6, 8, 16, 20, 24 and 48
  Patient-reported Chronic GVHD-specific Measures are defined by the National Institutes of Health (NIH) Consensus Development Project Criteria (2014).
Clinician-Assessed Global Rating/Scale | Week 0, 2, 4, 6, 8, 16, 20, 24 and 48
  Global Rating(0~3)/Scale(0~10) of clinician-assessed chronic GVHD-specific measures are defined by the National Institutes of Health (NIH) Consensus Development Project Criteria (2014).
Failure-free Survival | Week 24 and 48
  Failure-free survival, defined as absence of relapse, death and addition of new treatment, survival free of impairment, or reduction in steroid dosing that do not rely on direct assessment of organ responses.

CONTACTS AND LOCATIONS:
Locations (11):
- South Korea (11):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Inha University Hospital, Incheon
  - Seoul National University Seoul, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No